CLINICAL TRIAL: NCT03827070
Title: New Method of Treatment for Thoracoscopy or Bronchoscopy by Suspension of Fine Powder of Talcum and Afatinib is Used in Patients With Positive Mutation of EGFR in Non-Small Cell Lung Carcinoma (NSCLC)
Brief Title: Dry Pleurodesis With Talcum and Afatinib is Used to Treat Patients With Non-Small Cell Lung Carcinoma
Acronym: DPTA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center Trials & Treatment Europe (Network)
Collaborators: Center Trials & Treatment (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9TJJ425H1D
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Afatinib; Talcum powder; Thoracoscopy; Pleurodesis; BIBW2992
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Talc

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talcum powder & Afatinib (Experimental): Talcum powder 4 g + Afatinib 0,4 g. Is entered once
  Interventions: Drug: Afatinib; Drug: Talcum powder

INTERVENTIONS:
Drug: Afatinib — Used Afatinib particles of which had an average size of 22 μm and a volume concentration of small particles (<5 μm) - only 19%
  Other Names: BIBW2992
Drug: Talcum powder — Used Talcum powder particles of which had an average size of 24.5 μm and a volume concentration of small particles (<5 μm) - only 11%
  Other Names: Talc

SUMMARY:
In non-small cell lung cancer and metastases in the pleural cavity, pathological effusion is formed.

Currently, the most common and effective method of obliteration of the pleural cavity is pleurodesis with talcum powder.

Talc, when it surface of the pleura, causes chemical inflammation that leads to the soldering of the lungs and chest wall. As a result, the liquid ceases to accumulate.

The addition of a therapeutic dose of afatinib to talc not only blocks effusion into the pleural cavity, but also reduces tumor and metastatic processes.

DETAILED DESCRIPTION:
The proposed procedure for dry pleurodesis consists of one stage.

Talc is introduced into the pleural cavity in several ways:

* Drainage - a tube is inserted into the pleural cavity through a puncture in the chest, and then a pasty talcum is delivered into the cavity, which spreads through the cavity during the change of the patient's body position.
* Talcum powder - under the control of thoracoscopy, dry talc is blown into the pleural cavity of the patient, which allows him to evenly distribute and significantly increases the effectiveness of the procedure.

In this Clinical Trial investigators will use the method of thoracoscopy - the blow in of talcum powder and therapeutic dose of Afatinib. Before injection, a suspension of talc and afatinib is subjected to the procedure of pharmaceutical mixing.

The operation is well tolerated by participants and lasts no more than 30 minutes. The effectiveness of the method is 90%.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer with positive mutation of EGFR verified
* Malignant pleural effusion
* Recurrent pleural effusion
* Complete lung expansion (> 80%) after puncture emptying confirmed by chest radiography.
* Karnofsky index > 50
* Agreed to participate in the study and sign an Informed Consent

Exclusion Criteria:

* Radiotherapy not earlier than 3 months before the pleurodesis procedure
* Previous surgeries on the same hemitorace
* Thrombocytopenia or coagulation disorders
* Trapped lung syndrome
* Patients with estimated life expectancy < 4-8 weeks
* Pleural or active systemic infection

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-07-21 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the procedure of dry pleurodesis through a thoracoscope | up to 90 days
  Evaluation of the effectiveness of the dry pleurodesis procedure in combination with talc and afatinib with the introduction of a powder suspension through a thoracoscope.
  The assessment is performed by CT (computed tomography) of each participant twice: 30 days from the day of the procedure and 90 days later.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Contact, Tbilisi, Georgia